CLINICAL TRIAL: NCT00603876
Title: Efficacy of Almonds Added to Chronic Statin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Janelle Ruisinger, PharmD, Clinical Associate Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU FY08 GRF; 10998
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Step 1 dietary counseling plus 100-110 grams of almonds daily
  Interventions: Dietary Supplement: Almonds
- 1 (No Intervention): Step 1 dietary counseling

INTERVENTIONS:
Dietary Supplement: Almonds — 100-110 grams (about 3/4 cupful)of almonds consumed daily for 28 days
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the effects of 100-110 grams of almonds (about ¾ cupful) daily on the lipoprotein profile when given to patients on a statin drug. The study will compare the effects on the lipoprotein profile to patients who eat almonds and those patients not eating almonds.

DETAILED DESCRIPTION:
The primary objectives of this study are to determine the changes in the lipid profile [LDL-C, HDL-C, triglycerides, total cholesterol], LDL-C particle size, and the emerging risk factor Lp(a) when 100-110 g of almonds daily are added to statin therapy. Also, all subjects will receive Step I dietary counseling.

ELIGIBILITY:
Inclusion Criteria:

* Stable on current statin regimen for at least 8 weeks with plans to continue on the same dose while participating in the study
* Male or non-pregnant female - Women are eligible if they are surgically sterile or postmenopausal not using hormone replacement therapy (HRT) or using a stable, consistent does of HRT with intentions to continue therapy throughout the course of the study. Females of childbearing potential are eligible if using an effective form or contraception and intention to continue use through the study
* Mentally competent to understand study
* Speak and read English
* Able to maintain current medication regimen throughout study duration

Exclusion Criteria:

* LDL-C levels <70mg/dL
* Currently taking lipid-lowering agents other than statins including niacin, bile-acid sequestrants, ezetimibe, fibrates, high-dose Omega-3 fish oils (>1500mg of combined EPA/DHA daily) and policosanol
* Adherence to specialized diet regimes, i.e., multiple food allergies or nut allergy, vegetarian, macrobiotic, fad or popular diets, taking diet pills, etc.
* Already consuming nuts more than twice a week
* Active liver disease or a history of liver disease
* Chronic disease involving, hepatic, renal or coronary artery disease
* Currently taking systemic steroidal drugs
* Dependence on alcohol (> 10 drinks per week) or illicit drugs
* Participation in any other clinical trial within the last 30 days
* Engages in moderate intensity exercise for > 30 minutes each day
* Presence of any medical or psychological condition that in the opinion of the investigator will compromise safe subject participation for the duration of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measure of lipid panel including subfractions and Lp(a) and almond adherence | Once a month

SECONDARY OUTCOMES:
Measurement of height, weight, waist circumference, blood pressure and physical activity | Once a month

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Ruisinger, Pharm.D., Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - KU MedWest, Shawnee, Kansas

REFERENCES:
- [Derived] Ruisinger JF, Gibson CA, Backes JM, Smith BK, Sullivan DK, Moriarty PM, Kris-Etherton P. Statins and almonds to lower lipoproteins (the STALL Study). J Clin Lipidol. 2015 Jan-Feb;9(1):58-64. doi: 10.1016/j.jacl.2014.10.001. Epub 2014 Oct 13. PMID 25670361